CLINICAL TRIAL: NCT05742867
Title: Patient Preferences of Treatment for the Patients Suffering From Muscle-invasive Urothelial Carcinoma of Bladder Following Radical Cystectomy in Japan
Brief Title: A Study to Evaluate Treatment Preferences for Japanese Participants With Muscle-invasive Urothelial Carcinoma of the Bladder
Acronym: SNUGGLE
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-6M4
Record Dates: First submitted 2023-02-01; First posted 2023-02-24 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort 1: High-risk Muscle-Invasive Bladder Cancer (MIBC) participants following radical cystectomy

SUMMARY:
The main purpose of this study is to identify important treatment attributes for post-radical cystectomy (RC) treatment for participants with MIBC (Muscle-Invasive Bladder Cancer) and assess the relative importance of treatment attributes for post-RC treatment in Japan.

ELIGIBILITY:
Inclusion Criteria:

* Must reside in Japan and able to speak/read Japanese for the interview/survey
* Must have a clinical diagnosis of Muscle-invasive bladder cancer (MIBC):

  * ypT2-ypT4a or ypN+ MIBC, with prior neoadjuvant cisplatin chemotherapy and underwent radical cystectomy
  * pT3-pT4a or pN+ MIBC, without prior neoadjuvant cisplatin chemotherapy and underwent radical cystectomy
* Must not have received any treatment related to MIBC after radical cystectomy

Exclusion Criteria:

* Determined by the physician as being unsuitable for the study (e.g. having any clinically significant psychiatric disorder, cognitive impairment, or having difficulty with communicating in Japanese)
* Confirmed diagnosis of other primary cancers at the time of obtaining consent
* Current participation in a MIBC clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population is composed of 115 Japanese participants, 18 years and older, with muscle-invasive urothelial carcinoma of the bladder following radical cystectomy.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 1 year after radical cystectomy
  Median overall survival (years)
5-year survival rate | Up to 1 year after radical cystectomy
  Defined as the percentage of patients that are alive after 5 years
Disease-free survival (DFS) | Up to 1 year after radical cystectomy
  Median disease-free survival (year)
Probability of side effect-related treatment discontinuation | Up to 1 year after radical cystectomy
  Defined as the percent likelihood that a patient will stop treatment due to a side effect
Number of participants who experience treatment side effects | Up to 1 year after radical cystectomy
  Defined as the percentage of participants who experience nausea, diarrhea, fatigue, skin-related side effects (e.g. pruritus, rash), endocrine system-related side effects (e.g. hypothyroidism), anemia, alopecia, reduced renal function, cardiac impairment, leukopenia, neutropenia, and thrombocytopenia due to treatment
Overall severity of side effects | Up to 1 year after radical cystectomy
  Defined as the severity of side effects categorized as "None", "mild-to-moderate", or "severe"
Treatment Convenience | Up to 1 year after radical cystectomy
  Defined as the route of administration and frequency of administration per day or week (Infusions once every week, 2 weeks, or 4 weeks)
Treatment duration | Up to 1 year after radical cystectomy
  Defined as the total duration for continuous administration of treatment categorized as 2 months, 4 months, or 1 year
Hospitalization | Up to 1 year after radical cystectomy
  Defined as the length of hospitalization required for administration of treatment categorized as 0 days (no hospitalization required for administration of treatment), 1 week, or more than 1 week
Frequency of outpatient consultations | Up to 1 year after radical cystectomy
  Defined as the number of outpatient consultations required for treatment administration and monitoring categorized as every 2 weeks, 4 weeks, or 3 months
Annual treatment costs | Up to 1 year after radical cystectomy
  Defined as the annual out-of-pocket treatment costs, categorized as 10,000, 300,000, or 650,000 JPY

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Morrisville, North Carolina, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome